CLINICAL TRIAL: NCT02833675
Title: Determination of Specific Biomarkers of Angioneurotic Crisis
Acronym: BIOBRAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC12.210
Record Dates: First submitted 2016-06-28; First posted 2016-07-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Angioedema
Keywords: angioedema; C1Inhibitor; bradykinin; Histamin
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- bradykinin angioedema: Hereditary angioedema with or without C1Inhibitor Drug induced angiodema
- Histaminergic angioedema: Allergic and non allergic angioedema
- Control group: Patients with abdominal pain

SUMMARY:
Diagnosis of angioedema (AE) is difficult especially in emergency room. Two forms should be evoked: histaminic AE (allergic or not, which represent 95% of cases) and bradykinic AE (hereditary or acquired deficiency, with or without C1 Inhibitor) rarer but with more severe prognosis. The distinction is based on clinical features (spontaneous crisis duration, presence of concomitant hives, atopic history...). Sometimes it could be difficult to make the difference. Nowadays, there is no biological marker of the crisis. The search for biomarkers could improve the diagnostic and therapeutic management of AE. Previous work has identified targets: D-dimer, C4, and VE-cadherin. We wanted to know the sensitivity and specificity of these markers.

We conducted a prospective study evaluating the D-dimer assays, complement and VE-cadherin during an episode of AE. Three groups of patients were tested: bradykinic AE (peripheral or abdominal attacks), histaminic AE, and abdominal pain (non-bradykinic and non-histaminic etiology) at the time (day 0) and at distance from the crisis (D7).

ELIGIBILITY:
Inclusion Criteria:

* Histaminergic or bradykinin angioedema
* Abdominal pain

Exclusion Criteria:

* children < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bradykinin and histaminergic angioedema or with abdominal pain
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
VE CADHERIN SENSITIVITY AND SPECIFICITY | 7 DAYS

SECONDARY OUTCOMES:
D-DIMERS SENSITIVITY AND SPECIFICITY | 7 DAYS
C1INHIBITOR | 7 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa espin, Study Chair — grenbole university hospital
Locations (1):
- Grenoble university hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bowen T, Cicardi M, Farkas H, Bork K, Longhurst HJ, Zuraw B, Aygoeren-Pursun E, Craig T, Binkley K, Hebert J, Ritchie B, Bouillet L, Betschel S, Cogar D, Dean J, Devaraj R, Hamed A, Kamra P, Keith PK, Lacuesta G, Leith E, Lyons H, Mace S, Mako B, Neurath D, Poon MC, Rivard GE, Schellenberg R, Rowan D, Rowe A, Stark D, Sur S, Tsai E, Warrington R, Waserman S, Ameratunga R, Bernstein J, Bjorkander J, Brosz K, Brosz J, Bygum A, Caballero T, Frank M, Fust G, Harmat G, Kanani A, Kreuz W, Levi M, Li H, Martinez-Saguer I, Moldovan D, Nagy I, Nielsen EW, Nordenfelt P, Reshef A, Rusicke E, Smith-Foltz S, Spath P, Varga L, Xiang ZY. 2010 International consensus algorithm for the diagnosis, therapy and management of hereditary angioedema. Allergy Asthma Clin Immunol. 2010 Jul 28;6(1):24. doi: 10.1186/1710-1492-6-24. PMID 20667127
- [Background] Bluestein HM, Hoover TA, Banerji AS, Camargo CA Jr, Reshef A, Herscu P. Angiotensin-converting enzyme inhibitor-induced angioedema in a community hospital emergency department. Ann Allergy Asthma Immunol. 2009 Dec;103(6):502-7. doi: 10.1016/S1081-1206(10)60267-0. PMID 20084844
- [Background] Bork K, Siedlecki K, Bosch S, Schopf RE, Kreuz W. Asphyxiation by laryngeal edema in patients with hereditary angioedema. Mayo Clin Proc. 2000 Apr;75(4):349-54. doi: 10.4065/75.4.349. PMID 10761488
- [Background] Agostoni A, Cicardi M. Hereditary and acquired C1-inhibitor deficiency: biological and clinical characteristics in 235 patients. Medicine (Baltimore). 1992 Jul;71(4):206-15. doi: 10.1097/00005792-199207000-00003. PMID 1518394
- [Background] Cugno M, Zanichelli A, Bellatorre AG, Griffini S, Cicardi M. Plasma biomarkers of acute attacks in patients with angioedema due to C1-inhibitor deficiency. Allergy. 2009 Feb;64(2):254-7. doi: 10.1111/j.1398-9995.2008.01859.x. Epub 2008 Dec 4. PMID 19076541
- [Background] Bouillet L, Mannic T, Arboleas M, Subileau M, Massot C, Drouet C, Huber P, Vilgrain I. Hereditary angioedema: key role for kallikrein and bradykinin in vascular endothelial-cadherin cleavage and edema formation. J Allergy Clin Immunol. 2011 Jul;128(1):232-4. doi: 10.1016/j.jaci.2011.02.017. Epub 2011 Mar 24. No abstract available. PMID 21439626
- [Background] Grattan C, Powell S, Humphreys F; British Association of Dermatologists. Management and diagnostic guidelines for urticaria and angio-oedema. Br J Dermatol. 2001 Apr;144(4):708-14. doi: 10.1046/j.1365-2133.2001.04175.x. PMID 11298527
- [Background] Zingale LC, Beltrami L, Zanichelli A, Maggioni L, Pappalardo E, Cicardi B, Cicardi M. Angioedema without urticaria: a large clinical survey. CMAJ. 2006 Oct 24;175(9):1065-70. doi: 10.1503/cmaj.060535. PMID 17060655
- [Background] Temino VM, Peebles RS Jr. The spectrum and treatment of angioedema. Am J Med. 2008 Apr;121(4):282-6. doi: 10.1016/j.amjmed.2007.09.024. PMID 18374684
- [Background] Davis AE 3rd. The pathophysiology of hereditary angioedema. Clin Immunol. 2005 Jan;114(1):3-9. doi: 10.1016/j.clim.2004.05.007. PMID 15596403
- [Background] Moreau ME, Garbacki N, Molinaro G, Brown NJ, Marceau F, Adam A. The kallikrein-kinin system: current and future pharmacological targets. J Pharmacol Sci. 2005 Sep;99(1):6-38. doi: 10.1254/jphs.srj05001x. PMID 16177542
- [Background] Bas M, Adams V, Suvorava T, Niehues T, Hoffmann TK, Kojda G. Nonallergic angioedema: role of bradykinin. Allergy. 2007 Aug;62(8):842-56. doi: 10.1111/j.1398-9995.2007.01427.x. PMID 17620062
- [Background] Lumry WR, Castaldo AJ, Vernon MK, Blaustein MB, Wilson DA, Horn PT. The humanistic burden of hereditary angioedema: Impact on health-related quality of life, productivity, and depression. Allergy Asthma Proc. 2010 Sep-Oct;31(5):407-14. doi: 10.2500/aap.2010.31.3394. PMID 20929608
- [Background] Bygum A. Hereditary angio-oedema in Denmark: a nationwide survey. Br J Dermatol. 2009 Nov;161(5):1153-8. doi: 10.1111/j.1365-2133.2009.09366.x. Epub 2009 Jun 22. PMID 19709101
- [Background] Bork K, Meng G, Staubach P, Hardt J. Hereditary angioedema: new findings concerning symptoms, affected organs, and course. Am J Med. 2006 Mar;119(3):267-74. doi: 10.1016/j.amjmed.2005.09.064. PMID 16490473
- [Background] Bork K, Staubach P, Eckardt AJ, Hardt J. Symptoms, course, and complications of abdominal attacks in hereditary angioedema due to C1 inhibitor deficiency. Am J Gastroenterol. 2006 Mar;101(3):619-27. doi: 10.1111/j.1572-0241.2006.00492.x. Epub 2006 Feb 8. PMID 16464219
- [Background] Craig TJ, Wasserman RL, Levy RJ, Bewtra AK, Schneider L, Packer F, Yang WH, Keinecke HO, Kiessling PC. Prospective study of rapid relief provided by C1 esterase inhibitor in emergency treatment of acute laryngeal attacks in hereditary angioedema. J Clin Immunol. 2010 Nov;30(6):823-9. doi: 10.1007/s10875-010-9442-1. Epub 2010 Jul 16. PMID 20635155
- [Background] Cicardi M, Banerji A, Bracho F, Malbran A, Rosenkranz B, Riedl M, Bork K, Lumry W, Aberer W, Bier H, Bas M, Greve J, Hoffmann TK, Farkas H, Reshef A, Ritchie B, Yang W, Grabbe J, Kivity S, Kreuz W, Levy RJ, Luger T, Obtulowicz K, Schmid-Grendelmeier P, Bull C, Sitkauskiene B, Smith WB, Toubi E, Werner S, Anne S, Bjorkander J, Bouillet L, Cillari E, Hurewitz D, Jacobson KW, Katelaris CH, Maurer M, Merk H, Bernstein JA, Feighery C, Floccard B, Gleich G, Hebert J, Kaatz M, Keith P, Kirkpatrick CH, Langton D, Martin L, Pichler C, Resnick D, Wombolt D, Fernandez Romero DS, Zanichelli A, Arcoleo F, Knolle J, Kravec I, Dong L, Zimmermann J, Rosen K, Fan WT. Icatibant, a new bradykinin-receptor antagonist, in hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):532-41. doi: 10.1056/NEJMoa0906393. PMID 20818888
- [Background] Nussberger J, Cugno M, Cicardi M, Agostoni A. Local bradykinin generation in hereditary angioedema. J Allergy Clin Immunol. 1999 Dec;104(6):1321-2. doi: 10.1016/s0091-6749(99)70030-8. No abstract available. PMID 10589018
- [Background] Wallez Y, Vilgrain I, Huber P. Angiogenesis: the VE-cadherin switch. Trends Cardiovasc Med. 2006 Feb;16(2):55-9. doi: 10.1016/j.tcm.2005.11.008. PMID 16473763
- [Background] Hermant B, Bibert S, Concord E, Dublet B, Weidenhaupt M, Vernet T, Gulino-Debrac D. Identification of proteases involved in the proteolysis of vascular endothelium cadherin during neutrophil transmigration. J Biol Chem. 2003 Apr 18;278(16):14002-12. doi: 10.1074/jbc.M300351200. Epub 2003 Feb 12. PMID 12584200
- [Background] Lambeng N, Wallez Y, Rampon C, Cand F, Christe G, Gulino-Debrac D, Vilgrain I, Huber P. Vascular endothelial-cadherin tyrosine phosphorylation in angiogenic and quiescent adult tissues. Circ Res. 2005 Feb 18;96(3):384-91. doi: 10.1161/01.RES.0000156652.99586.9f. Epub 2005 Jan 20. PMID 15662029
- [Background] Brevet: w/o 2008 062314 circulating ve-cadherin as a predictive marker of sensitivity or resistance to anti-tumoral treatment, and improved method for the detection of soluble proteins.